CLINICAL TRIAL: NCT01756443
Title: Sciatic Nerve Block for Ankle/Foot Surgeries. A Comparison Between a Premixed Solution of Lidocaine Plus Bupivacaine and Consecutive Infiltration of Lidocaine and Bupivacaine. A Double Blinded Randomised Controlled Prospective Study
Brief Title: Sciatic Nerve Block for Ankle/Foot Surgeries. A Comparison Between a Premixed Solution of Lidocaine Plus Bupivacaine and Consecutive Infiltration of Lidocaine and Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, DR. Jassim Rauf, Clinical Research/ Peripheral Nerve Blocks Fellow., Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JR-786-GI; SQ-PM-40
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Open Reduction Internal Fixation(ORIF) of Lateral Malleolus
Keywords: sciatic nerve block; ORIF lateral malleolus; sequential injection; premixed injection; local anaesthetics
MeSH Terms: interventions — Lidocaine; Epinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premixed group (Active Comparator): Patients will receive sciatic nerve block with premixed 7.5 mls of 2% lidocaine/adrenaline and 7.5 mls of 0.5% bupivacaine followed by an interval of 90 seconds with an injection of same amount of both drugs.
  Interventions: Drug: 2% lidocaine/adrenaline and 0.5% bupivacaine
- Sequential Group (Experimental): Patients will receive a sciatic nerve block with 15 mls of 2% lidocaine/adrenaline followed by an interval of 90 seconds with 15 mls of 0.5% bupivacaine.
  Interventions: Drug: 2% lidocaine/adrenaline and 0.5% bupivacaine

INTERVENTIONS:
Drug: 2% lidocaine/adrenaline and 0.5% bupivacaine

SUMMARY:
Regional anaesthesia has become the cornerstone of multimodal analgesia. With the advent of ultrasound guided nerve blocks regional anaesthesia has achieved both greater efficacy and a better safety profile as the injection of local anaesthetic is performed under direct vision. This has allowed a reduction of the amount of local anaesthetic injected as compared to peripheral nerve stimulation technique . Blockade of sciatic nerve combined with saphenous nerve provides anaesthesia and analgesia for ankle/foot surgeries. Various combinations of local anaesthetics have been used to provide optimal blockade . A mixture of lidocaine with a long acting local anaesthetic is commonly used. This provides a rapid onset of blockade, but of a consistently shorter duration compared to a long acting local anaesthetic alone. We hypothesize that sequential perineural injection of lidocaine and bupivacaine provides similar onset but a longer duration of sensory block compared to the same dose and volume of local anaesthetic mixed in advance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA 1 - 3 status
* scheduled to undergo semi-elective ankle/foot surgery under regional anaesthesia +/- sedation/opioid free general anaesthesia will be recruited

Exclusion Criteria:

* Patients having surgery on the medial aspect of the ankle/ foot
* allergy to local anaesthetics
* coagulopathy
* malignancy or infection in the popliteal area
* significant peripheral neuropathy
* neurologic disorder of the lower extremity
* any other contraindication to sciatic nerve block
* pregnancy
* history of alcohol or drug dependency/abuse (defined as >40 IU/week)
* a history of significant cognitive or psychiatric disorder that may affect patient assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia/duration of block | 24 hours

SECONDARY OUTCOMES:
onset of block | 40 minutes
  the block will be assessed every 5 minutes from the time of needle withdrawal till complete loss of sensation to touch.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Iohom, MB, Phd, Principal Investigator — Cork University Hospital, Cork, Ireland
Locations (1):
- Cork University Hospital, Cork, Ireland